CLINICAL TRIAL: NCT03679611
Title: Impact of Sugammadex vs. Neostigmine Reversal on Post-Operative Recovery And Postoperative Complications In Patients With Obstructive Sleep Apnea Undergoing Bariatric Surgery: A Double-Blind, Randomized Controlled Trial
Brief Title: Impact of Sugammadex vs. Neostigmine Reversal on Post-Operative Recovery and Complications
Acronym: Sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Canada Inc. (Industry)
Responsible Party: Principal Investigator, Jean Wong, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-5629
Record Dates: First submitted 2018-09-13; First posted 2018-09-20 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Recovery time; reversal of neuromuscular blockers (NMB); obstructive sleep apnea; morbid obesity; bariatric surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity, Morbid | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Intervention Model Description: This study is a prospective, double-blinded randomized controlled superiority trial with two parallel groups. Randomization will be performed with a 1:1 allocation into reversal of neuromuscular blocking drugs (NMBD) with sugammadex or neostigmine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study investigators, research coordinator, patients, surgeons, anesthesiologists, health care personnel will be blinded to the treatment arm allocation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): Interventional Arm will receive sugammadex sodium 2 mg/kg actual body weight, At the end of surgery Sugammadex will be administered when the TOF reveals at least 2 responses
  Interventions: Drug: Sugammadex Sodium
- Standard drug Arm (Active Comparator): standard drug Arm will receive neostigmine 2.5 mg and glycopyrrolate 0.4 mg, At the end of surgery neostigmine and glycopyrrolate will be administered when the TOF reveals at least 2 responses
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex Sodium — Sugammadex is a FDA approved newer NMBD reversal agent. But does not use in standard of care in most of institutions This study is designed to compare the impact of reversal of neuromuscular blockade with sugammadex vs. neostigmine on discharge time from the operating room in obese patients with OSA undergoing bariatric surgery
  Other Names: Bridion
  Arms: Interventional Arm
Drug: Neostigmine — neostigmine is a FDA approved NMBD reversal drug, uses as standard care drug in most of the institutions. neostigmine use as active comparator to compare with investigational drug Sugammadex in the study.
  Other Names: prostigmin
  Arms: Standard drug Arm

SUMMARY:
Sugammadex or neostigmine are given at the end of the surgery to reverse neuro muscular blocking drugs (NMBD). This study will evaluate whether reversal of NMBD with sugammadex is associated with faster recovery than neostigmine resulting in faster discharge from the operating room (OR) in obese patients with OSA undergoing bariatric surgery. Half of the patients in the study will receive sugammadex and the other half of the patients will receive neostigmine.

DETAILED DESCRIPTION:
Sugammadex and neostigmine are NMBD reversal agents. Neostigmine - an anticholinesterase is given to reverse NMBD; however reversal of NMBD with neostigmine may be associated with residual neuromuscular blockade in up to 64% patients postoperatively in the post anesthesia care unit. Even mild degrees of residual neuromuscular blockade can have serious clinical consequences in the postoperative period. The severity of OSA often worsens after surgery and patients with OSA are at increased risk for early respiratory complications after extubating and in the PACU. Morbid obesity is associated with critical respiratory complications in patients with OSA.

Sugammadex is a newer NMBD reversal agent that rapidly and completely reverses rocuronium. It is a modified gamma cyclodextrin that forms a complex with the neuromuscular blocking agent rocuronium. It reduces the amount of neuromuscular blocking agent available to bind to nicotinic cholinergic receptors in the neuromuscular junction. It has been shown to more rapidly reverse residual neuromuscular blockade than neostigmine in obese patients without obstructive sleep apnea (OSA).

This study will evaluate whether reversal of NMBD with sugammadex is associated with faster recovery than neostigmine resulting in faster discharge from the operating room (OR) in obese patients with OSA undergoing bariatric surgery. Half of the patients in the study will receive sugammadex and other half of the patients will receive neostigmine

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosed Obstructive Sleep Apnea patients by polysomnography
* Scheduled elective bariatric surgery

Exclusion Criteria:

* Age<18 years old
* Allergy to rocuronium
* Allergy to sugammadex
* Allergy to neostigmine
* Malignant hyperthermia
* Hepatic insufficiency
* Renal insufficiency
* Neuromuscular Disease
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, Principal Investigator — University Health Network, Toronto Western Hospital
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Research study results will be presented for publication in peer reviewed journals by the protocol.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 patients were enrolled from January 14, 2019 to October 26, 2021. Study coordinators screened 237 patients for eligibility in the pre-operative and bariatric clinics at Toronto Western Hospital, University Health Network- a Bariatric Centre of Excellence located in Toronto, Ontario, Canada. Consenting patients were ≥18 years with OSA diagnosed by polysomnography for elective bariatric surgery under general anesthesia. Randomization was 1:1 into 2 groups of sugammadex vs. neostigmine.
Pre-assignment Details: A total of 237 patients were screened for eligibility in our study. 108 were excluded for not meeting study criteria. 9 were excluded for reasons like a hold on surgeries due to the coronavirus disease (COVID-19) pandemic or cancellations, unavailability of investigators on scheduled surgery days, etc. 120 patients were enrolled on the study and were subsequently randomized 1:1 into 2 groups of 60 patients each, given the study drug, and followed-up as per the study protocol.
Groups:
- Interventional Arm: Interventional Arm will receive sugammadex sodium 2 mg/kg actual body weight, At the end of surgery Sugammadex will be administered when the TOF reveals at least 2 responses
  Sugammadex Sodium: Sugammadex is an FDA approved newer neuromuscular blocking drug (NMBD) reversal agent. But does not use in standard of care in most of institutions This study is designed to compare the impact of reversal of neuromuscular blockade with sugammadex vs. neostigmine on discharge time from the operating room in obese patients with OSA undergoing bariatric surgery
Period: Overall Study
Arm/Group | Interventional Arm | Standard Drug Arm
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study population were morbidly obese adult (≥18 years) patients with OSA diagnosed by polysomnography for elective bariatric surgery under general anesthesia at Toronto Western Hospital- University Health Network, who were able to give consent. They were randomized 1:1 for reversal of NMBDs with sugammadex or neostigmine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional Arm | Standard Drug Arm | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 49.50 [43.75 to 54.00] | 51.00 [42.75 to 55.25] | 50.50 [43.00 to 55.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 15 | 17 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Time to Discharge From Operating Room
Description: The time from study drug administration to discharge from operating room (OR).
Time Frame: 15 minutes
Population: Same as baseline
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Interventional Arm | Standard Drug Arm
Number analyzed (Participants) | 60 | 60
Minutes | 13.0 [10.0 to 15.0] | 13.5 [11.0 to 15.0]

2. Secondary Outcome: Time the Patient Open Eyes to Command
Description: Time from study drug administration to the patient open eyes to command.
Time Frame: 15 minutes
Population: Same as baseline
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Interventional Arm | Standard Drug Arm
Number analyzed (Participants) | 60 | 60
Minutes | 6.00 [4.00 to 10.00] | 7.00 [4.00 to 10.00]

3. Other Pre Specified Outcome: Time to Extubation
Description: Time from study drug administration to extubation
Time Frame: 15 minutes
Population: Same as baseline
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Interventional Arm | Standard Drug Arm
Number analyzed (Participants) | 60 | 60
Minutes | 7.00 [5.00 to 11.00] | 8.00 [6.00 to 11.00]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected when available through the course of study completion for each participant, an average of 1 day.
Description: Standard definitions were used by the study for adverse events.
Arm/Group | Interventional Arm | Standard Drug Arm
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=60) | Standard Drug Arm (N=60)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Spontaneous resolution/self limiting. Less than 24 hours. Assessed as mild and unrelated.
Cellulitis left leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Resolved. 10 days. Assessed as moderate and unrelated

LIMITATIONS AND CAVEATS:
1. . USFDA recommends neostigmine 0.03 mg/kg to 0.07 mg/kg. We used 2.5 mg for NMBD reversal. A less-than-recommended dose being used in our patients. However, providers had the option of giving a supplemental dose of neostigmine or sugammadex if they felt it was clinically indicated, with a very low rate of redosing
2. . Lack of continuous quantitative neuromuscular monitoring and ability to detect residual NMBD at the time of extubating
3. . Conservative use of muscle relaxants by our providers

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03679611/Prot_SAP_000.pdf